CLINICAL TRIAL: NCT05926323
Title: Anesthesia Quality Control Indicators of 6 Provinces in Central China
Status: Withdrawn | Type: Observational
Sponsor: Shanglong Yao (Other)
Responsible Party: Sponsor-Investigator, Shanglong Yao, Professor; Director of Hubei Provincial Anesthesia Quality Control Center, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: AQCICC
Record Dates: First submitted 2023-06-18; First posted 2023-07-03 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia-related Quality Control Indicators; Anesthesia-related Adverse Events

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators are aimed to evaluate the anaesthesia-related quality control indicators and adverse events, in terms of its incidence, changes, causes, risk factors and preventability in Central China, using a series of annual surveys.

DETAILED DESCRIPTION:
The investigators prospectively collected information on patient, surgical, anaesthesia, and hospital characteristics for all anaesthesia procedures performed in all certified facilities in Central China. All available data of patients who had anaesthesia were gathered monthly from anaesthesia quality control groups that provide services to all certified facilities and were reviewed.

All anaesthesia-related adverse events were scrutinized consecutively to determine their root causes and preventability. The incidence and patterns of anaesthesia-related quality control indicators and adverse events were analysed.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing anesthesia

Exclusion Criteria:

Those with a miss-reporting rate higher than 5%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
number of anesthesia per anesthesiologist | through study completion, an average of 1 year
proportion of patients of different American Society of Anesthesiologists physical status (ASAPS) | through study completion, an average of 1 year
proportion of emergency non selective anesthesia | through study completion, an average of 1 year
proportion of various anesthesia methods | through study completion, an average of 1 year
proportion of intraoperative autologous blood transfusion | through study completion, an average of 1 year
cancellation of operations after the anesthesia | through study completion, an average of 1 year
delayed transfer from the post-anesthesia care unit (PACU) | through study completion, an average of 1 year
hypothermia in the PACU | through study completion, an average of 1 year
unplanned transfer to intensive care unit (ICU) | through study completion, an average of 1 year
unplanned secondary tracheal intubation | through study completion, an average of 1 year
anesthesia-related death within 24 hours of anesthesia | through study completion, an average of 1 year
  Anesthesia-related deaths were diagnosed and reported timely by the data-quality-control staffs at all AQCC certified facilities, according to the time and code of death.
  Time: within 24 h of anesthesia induction Code: International Classification of Diseases, 10th Revision for medical conditions related to anesthesia or anesthetics was grouped into four categories: (1) complications of anesthesia during labor (24 hours after anesthesia); (2) overdose of anesthetics for surgical purposes; (3) adverse effects of anesthetics in therapeutic use; and (4) other complications of anesthesia in surgical and medical care
cardiac arrest within 24 hours of anesthesia | through study completion, an average of 1 year
severe anaphylaxis during anesthesia | through study completion, an average of 1 year
severe neurological complications after intraspinal anesthesia | through study completion, an average of 1 year
serious complications of central venipuncture | through study completion, an average of 1 year
hoarseness after tracheal catheter extubation | through study completion, an average of 1 year
coma after anesthesia | through study completion, an average of 1 year